CLINICAL TRIAL: NCT06238765
Title: CorEvitas International Adolescent Atopic Dermatitis (AD) Drug Safety and Effectiveness Registry
Status: Recruiting | Type: Observational
Sponsor: CorEvitas (Network)
Responsible Party: Sponsor
Other Study IDs: CorEvitas-AD-555
Record Dates: First submitted 2024-01-16; First posted 2024-02-02 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective observational registry for an adolescent cohort with AD under the care of a dermatology provider. Approximately 1500 subjects and 75 clinical sites in North America and select European countries will be recruited to participate with no defined upper limit for either target.

DETAILED DESCRIPTION:
The objective of the registry is to create a cohort of adolescent subjects with AD to evaluate the long-term safety and effectiveness of AD treatments. Data collected will be used to better characterize the natural history of the disease and to extensively evaluate the effectiveness and safety of medications approved for the treatment of AD to support ongoing risk-benefit evaluation by drug manufacturers and regulators. Further, data collected will inform clinical decision making by patients and treating providers. This will be done through standardized data collection including validated instruments for patient-reported outcomes (PROs) and clinician-reported outcomes (ClinROs), the active evaluation of prevalent and incident comorbidities and adverse events, and the recording of medication utilization patterns.

This provides an opportunity to evaluate other aspects of the disease and its treatment, including but not limited to clinical and drug cost-effectiveness, health care resource utilization, and subject adherence.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in this registry, an individual must meet all the following criteria:

  1. Has been diagnosed with moderate to severe atopic dermatitis by a dermatologist or a qualified dermatology practitioner.
  2. Is 12 - 15 years of age at the time of enrollment.
  3. Meets one of the following conditions at the time of enrollment:

     1. Has started taking a new Enrollment Eligible Medication within 6 months prior to the Enrollment visit. A new medication is a medication that the subject has never taken before.

        OR
     2. Is prescribed a new Enrollment Eligible Medication at the Enrollment visit. A new medication is a medication that the subject has never taken before.

        Exclusion Criteria:

        An individual who meets any of the following criteria will be excluded from participation in the registry:

  <!-- -->

  1. Is participating or planning to participate in a blinded clinical trial for an AD drug.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects can enroll as early as age 12 and will be followed until the age of 18; therefore, the maximum duration a subject can be enrolled is < 6 years.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-12-02 (Actual); Primary Completion 2099-12-31 (Estimated); Study Completion 2099-12-31 (Estimated)

PRIMARY OUTCOMES:
AD epidemiology, presentation, natural history, management, and outcomes | Through Study completion until the subject is 18 years
  The major clinical outcomes include an assessment of the epidemiology of Atopic Dermatitis; to better understand the presentation, natural history, management and outcomes.

SECONDARY OUTCOMES:
Percentage of patients with history of comorbidities | Time Frame: at registry enrollment
Physician reported: validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD | every 6 months until the subject is 18 years
  Score: 0-4, with high score indicating widespread of atopic dermatitis
Physician reported: Nail changes due to atopic dermatitis (graduated VAS) | every 6 months until the subject is 18 years
  Scale - 0 (Clear/Normal) to 100 (Severe Abnormalities). Lower numbers are for mild abnormalities in a few nails, higher numbers are for more severe changes in many nails
Atopic dermatitis body surface area (BSA) | every 6 months until the subject is 18 years
Eczema Area and Severity Index (EASI) (calculated) | every 6 months until the subject is 18 years
  The severity of each sign will be graded on a scale of 0 to 3: (0) None, (1) Mild, (2) Moderate, (3) Severe.
Physician reported : SCORing Atopic Dermatitis index (SCORAD) (calculated) | every 6 months until the subject is 18 years
  The severity of each sign will be graded on a scale of 0 to 3: (0) None, (1) Mild, (2) Moderate, (3) Severe. For the Overall Score [SCORAD], select a lesion that that is representative of the body and score using the same severity scale
Patient reported : Patient global assessments of disease control and severity | every 6 months until the subject is 18 years
  This determines the progression & severity of the disease
Physician reported : Pubertal Progression: Tanner Staging Assessment | Every six Months until a subject is 18 years or the subjects reaches stage 5 of the ranner stangins assessment
Patient reported: Patient Oriented Eczema Measure (POEM) | every 6 months until the subject is 18 years
Patient reported: Peak pruritus (itch) NRS | every 6 months until the subject is 18 years
Patient reported: Skin pain NRS | every 6 months until the subject is 18 years
Patient reported: Fatigue NRS | every 6 months until the subject is 18 years
Patient reported: Children's Dermatology Life Quality Index (CDLQI) | every 6 months until the subject is 18 years
Patient reported: Patient Health Questionnaire (PHQ-4) | every 6 months until the subject is 18 years
Patient reported: Atopic dermatitis control tool (ADCT) | every 6 months until the subject is 18 years
Patient reported: Asthma Control test | every 6 months until the subject is 18 years
Patient reported: Sleeplessness and average pruritus (itch) NRS (SCORAD) | 6 months until the subject is 18 years

CONTACTS AND LOCATIONS:
Locations (1):
- CorEvitas, LLC, Waltham, Massachusetts, United States